CLINICAL TRIAL: NCT05812872
Title: The Effect of Allograft, Toothgraft, Alloplast on Alveolar Ridge Preservation
Brief Title: Alveolar Ridge Preservation Using Different Bone Substitutes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIR092210
Record Dates: First submitted 2022-09-04; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Alveolar Ridge Enlargement
Keywords: Alveolar ridge preservation, Allograft, Toothgraft, Allopast
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alveolar ridge preservationwith tooth graft (Active Comparator): tooth graft
  Interventions: Drug: Toothgraft
- Alveolar ridge preservation with allograft (Active Comparator): Allograft
  Interventions: Drug: Allograft
- Alveolar ridge preservation with alloplast (Active Comparator): Beta Tri-Calcium phosphate
  Interventions: Drug: Alloplast

INTERVENTIONS:
Drug: Toothgraft — Particulate dentin
  Arms: Alveolar ridge preservationwith tooth graft
Drug: Allograft — Mineralized corticocancellous allograft
  Other Names: Mineralized corticocancellous allograft
  Arms: Alveolar ridge preservation with allograft
Drug: Alloplast — Beta tri-calcuim phosphate
  Other Names: Beta tri-calcuim phosphate
  Arms: Alveolar ridge preservation with alloplast

SUMMARY:
The primary objective of this study was to compare the efficacy of using allograft, autogenous tooth graft, and beta-tricalcium phosphate for alveolar ridge preservation (ARP) by examining the alveolar ridge height and width at baseline and 3 months after the ARP both clinically and radiographically. The secondary objective was to evaluate the quality of the newly formed bone using histomorphometric analysis.

DETAILED DESCRIPTION:
This randomized controlled clinical trial included thirty patients. ARP was performed using either Allograft (Allograft group n=10), Tooth graft (Toothgraft group n=10), and beta tri-calcium- phosphate (beta tri-calcium group n=10). Changes in alveolar ridge dimensions were evaluated clinically and radiographically using cone beam computed tomography at baseline and 3 months. Core bone biopsy samples were obtained 3 months post-extraction during implant placement for histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

1. seeking implant-based restorations after tooth extraction.
2. exhibited no evidence of any significant medical history, measured using Burket's Oral medicine health history questionnaire.
3. exhibited Type I and II sockets

Exclusion Criteria:

1. nonsmokers.
2. Pregnant and breast-feeding females
3. patients with known contraindications to dental implant surgery (e.g., increased bleeding tendency, history of treatments such as radiotherapy,

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Clinical assessment | 3 months
  Measure bone height loss in millimeter at baseline and after 3 months was measured using periodontal probe from the stent margin to the alveolar ridge crest at six points. In addition, Bone width loss was calculated by measuring alveolar ridge width buccopalatally in millimeter using a caliper clamp. The measurement was done perpendicular to the tangent of the dental arch at the mid-point of the extraction site approximately 4mm apical to the level of the marginal gingiva of the adjacent teeth.
Clinical assessment | 3 months
  Bone width loss was calculated by measuring alveolar ridge width buccopalatally in millimeter using a caliper clamp. The measurement was done perpendicular to the tangent of the dental arch at the mid-point of the extraction site approximately 4mm apical to the level of the marginal gingiva of the adjacent teeth.

SECONDARY OUTCOMES:
Radiographic assessment | 3 months
  Measuring loss in bone height in millimeters between baseline and after 3 months. Loss in bone height was calculated by measuring the distance from the alveolar crest both buccally and palatally to a fixed anatomical landmark. In addition,
Radiographic assessment | 3 months
  Loss in bone width was calculated by measuring distance from buccal alveolar crest to palatal alveolar crest in millimeter.

OTHER OUTCOMES:
Histological | 3 months
  Masson trichrome special stain was used to detect the area percentage of immature collagen and mature collagen at magnification 20X. The immature collagen appeared blue in color while areas with mature collagen appeared reddish in color
Histomorphometric analysis | 3 months
  Photomicrographs of 3 microscopic fields of each MT stained section, were captured at the original magnification of 20X using a digital camera(Canon EOS 650D) mounted on a light microscope(BX60,Olympus , Japan). The images were analyzed for obtaining the area percentage of mature and immature collagen of the newly formed bone using image J (1.41aNIH, USA)software

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine A Fouad, Ph.D, Principal Investigator — Ain Shams University; Suzan M Sarhan, Ph.D, Study Director — Ain Shams University; Hadeel M Gamal, Ph.D, Study Director — Ain Shams University; Basma A Abdelrahman, Ph.D, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt